CLINICAL TRIAL: NCT05414591
Title: A Phase 1 Clinical Trial to Compare and Evaluate the Safety and Pharmacokinetic Characteristics After Administration of DWP16001 Drug A and DWP16001 Drug B in Healthy Adult Volunteers
Brief Title: Pharmacokinetics and Safety Following Administration of DWP16001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWP16001105
Record Dates: First submitted 2022-06-08; First posted 2022-06-10 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence group A (Experimental): DWP16001 A mg 1T
  Interventions: Drug: DWP16001 drug A; Drug: DWP16001 drug B
- Sequence group B (Experimental): DWP16001 B mg 3T
  Interventions: Drug: DWP16001 drug A; Drug: DWP16001 drug B

INTERVENTIONS:
Drug: DWP16001 drug A — 1 tablet, Oral, once daily single dose
Drug: DWP16001 drug B — 3 tablet, Oral, once daily single dose

SUMMARY:
To compare and evaluate the safety and pharmacokinetic characteristics after administration of DWP16001 Drug A and DWP16001 Drug B in healthy adult volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers aged ≥ 19 years at screening
* Subjects with a body weight of ≥ 50.0 kg to ≤ 90.0 kg with a body mass index (BMI) of ≥ 18.0 kg/m2 and ≤ 30.0 kg/m2
* Subjects with no congenital or chronic disease that requires treatment, and no clinical symptoms or findings based on medical examination
* Subjects who are determined eligible to participate in this study based on results of laboratory tests, vital signs, physical examination etc at screening.

Exclusion Criteria:

* Current or history of clinically significant hepatic, renal, nervous, respiratory, endocrine, hemato-oncology, cardiovascular, urogenital, psychosis disorder
* Current or history of gastrointestinal disorders or prior history of gastrointestinal surgery that may affect safety and PK/PD assessment of the study drug
* Clinical laboratory test values are outside the accepted normal range at screening
* Other exclusive inclusion criteria, as defined in the protocol

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
AUC0_t of DWP16001 | 0-72 hours
  Area under the plasma concentration versus time curve
Cmax of DWP16001 | 0-72 hours
  Peak Plasma Concetration

SECONDARY OUTCOMES:
Tmax Tmax | 0-72 hours
  Time at Cmax Tmax
AUC of DWP16001 | 0-72 hours
  Area under the plasma concentration versus time curve
T 1/2 of DWP16001 | 0-72 hours
  half life of DWP16001
CL/F of DWP16001 | 0-72 hours
  Apparent total clearance of the drug from plasma after oral administration
Vd/F of DWP16001 | 0-72 hours
  Volume of distribution

CONTACTS AND LOCATIONS:
Locations (1):
- CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do, South Korea